CLINICAL TRIAL: NCT05504330
Title: Cognitive Decline and Underlying Mechanisms in Asymptomatic Intracranial Artery Stenosis Patients: A Cohort Study
Brief Title: Cognitive Decline and Underlying Mechanisms in Asymptomatic Intracranial Artery Stenosis Patients
Status: Recruiting | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab Anhui Medical University, PRC, Anhui Medical University
Other Study IDs: Anhui-AsIA-cohort
Record Dates: First submitted 2022-08-07; First posted 2022-08-17 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Asymptomatic Intracranial Stenosis; Cognitive Impairment; Cerebrovascular Event
Keywords: Asymptomatic Intracranial Stenosis patients; Cognitive Impairment; Cerebrovascular Event
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Aspirin; Clopidogrel; Atorvastatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and anticoagulant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient Group: Asymptomatic intracranial stenosis patients who receive standard medical treatment without stenting
  Interventions: Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin
- Healthy Control: Healthy control are free from intracranial stenosis

INTERVENTIONS:
Drug: Aspirin Tablet, Clopidogrel Bisulfate Tablets and Atorvastatin — First of all, ICAS patients were given health education to exhort them to reduce the risk factors of exposure to stroke and get rid of their unhealthy lifestyles. Secondly, for patients in need, standardize their dosage and course of treatment, mainly including antiplatelet drugs and statins. In addition, patients with diabetes and hypertension urge rational medication to control blood pressure and blood glucose level.
  Groups: Patient Group

SUMMARY:
The purpose of this study is to explore the mechanism of cognitive impairment in patients with asymptomatic intracranial atherosclerotic stenosis(ICAS),and to examine the natural history and the pathogenesis of asymptomatic ICAS.

DETAILED DESCRIPTION:
All participants underwent a medical evaluation that included routine laboratory studies before and after 1- and 2-years follow-up. Upon meeting the inclusion criteria and providing informed consent, each participant will complete a battery measure of neuropsychological tests, blood sample collection, and magnetic resonance imaging scan after enrollment and after 1- and 2-years follow-up.

About 100 participants were included in this study. A series of neuropsychological tests were obtained by a trained investigator to assess. The tests include the evaluation of global cognitive function and multiple individual cognitive domains. The various tasks and questionnaires to measure cognition function including Montreal Cognitive Assessment(MoCA), Mini Mental State Examination(MMSE), Chinese Auditory Verbal Learning Test(CAVLT), Digital Span Test(DST), Symbol digital modalities test(SDMT), Stroop color test(Stroop test), Color trail test(CTT), Rey-Osterrieth Complex Figure(ROCF), Judgment of Line Orientation (JoLO), Verbal Fluency Test(VFT), Boston Naming Test (BNT) , Lateralized attention network test(LANT) etc, at the same time, the investigators also pay attention to the evaluation of participants' emotions by Hamilton Anxiety Scale(HAMA),Hamilton Depression Scale(HAMD). Furthermore, the memory as the primary outcome measure, this study focused on the immediate memory, delayed memory and recognition memory of patients with asymptomatic ICAS. Blood sample will be collected for biological multiomics research. The patients will receive a magnetic resonance imaging scan in multi-modalities.

After 1 and 2 years follow-up,the participants will be interviewed to obtain the same assessments, blood sample and magnetic resonance imaging scan in multi-modalities as before.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with intracranial stenosis which was defined as stenosis of 50% or more in Intracranial segment of internal carotid artery(C6-C7) and middle cerebral artery (M1).
2. The degree of stenosis was measured by transcranial doppler, computed magnetic resonance angiography (MRA),tomography angiography (CTA) and digital subtraction angiography (DSA).

Exclusion Criteria:

1. History of stroke,transient ischemic attack,seizures or unexplained loss of consciousness.
2. Organic brain defects on MRI T1 or T2 images.
3. Any history or clinical signs of other severe psychiatric illnesses (like major depression,psychosis or obsessive compulsive disorder).
4. Implanted pacemaker,medication pump,vagal stimulator,deep brain stimulator. History of substance abuse within the last 6 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with intracranial stenosis which was defined as stenosis of 50% or more in Intracranial segment of internal carotid artery and middle cerebral artery (MCA) without history of stroke,transient ischemic attack,seizures or unexplained loss of consciousness.The degree of stenosis was measured by transcranial doppler, computed magnetic resonance angiography (MRA),tomography angiography (CTA) and digital subtraction angiography (DSA).
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The changes in Memory | baseline, 1 and 2 years after follow-up
  The changes in Memory function will constitute one of the main indicators of research results, which will be used to evaluate the follow-up results of the standard treatment regimen. The investigators will use the Chinese Auditory Verbal Learning Test (CAVLT) to evaluate the immediate, delayed and recognition memory of patients with asymptomatic ICAS to evaluate the immediate, delayed and recognition memory of patients with ICAS.
Occurrence of ischemic cerebrovascular events | baseline, 1 and 2 years after follow-up
  The changes in occurrence of ischemic cerebrovascular events constitute another major indicator of research result. The new responsible vascular cerebrovascular events during the follow-up period are also the clinical information the investigators pay attention to, including transient ischemic attack (TIA) and stroke.

SECONDARY OUTCOMES:
MoCA (Montreal Cognitive Assessment) | baseline, 1 and 2 years after follow-up
  The changes in MoCA will constitute the secondary research outcome. MoCA was based on clinical experience and reference to the MMSE cognitive items and scores, and the final version was finalized in November 2004. The investigators adopted a localized version (Mandarin version，includes 2 alternative versions) in line with the Chinese cultural background.It includes 11 inspection items in 8 cognitive fields, including visual structure skills, executive function, naming, attention and calculation, language, abstract thinking, memory, and orientation. With a total score of 30 or more than 26, it is normal. Anyone who has been education for less than 12 years will need to add one point to his final score. The final score of the higher the better.
MMSE (Mini Mental State Examination) | baseline, 1 and 2 years after follow-up
  The changes in MMSE will also constitute the secondary research outcome.The full name of MMSE is mini-mental state examination, and the scale consists of 30 subject, include the following seven aspects: time orientation, place orientation,immediate memory,attention and calculation,delay memory,language, visual space.One point is awarded for each question correctly answered during MMSE evaluation. If subject give the wrong answer or don't know answer he/she awarded 0 score, scope of scale score of 0 to 30 points. The higher the score, the better. In this study, the investigators suspect that scores would decrease after follow-up.
DST (Digital Span Test; Forward and Backward) | baseline, 1 and 2 years after follow-up
  The changes in DST will constitute the secondary research outcome. Digital span test (DST) was commonly used to evaluate attention ability and instantaneous memory ability. There are two types of test: forward(0-14) and backward(0-13).In the forward test, the subjects were asked to retell the the digits immediately after hearing it until they could not be repeated correctly.In backward test, the subjects were asked to repeat a set of numbers in reverse order until they could not be repeated correctly. The length of the last set of Numbers correctly repeated by the subjects was the final score, forward and backward are counted separately. The higher the score, the better. In this study, the investigators suspect that scores would decrease after follow-up.
SDMT (Symbol digital modalities test) | baseline, 1 and 2 years after follow-up
  The changes in The Symbol digital modalities test (SDMT) will constitute the secondary research outcome measure. The investigators intend to explore the cognitive processing speed of patients with SDMT, and evaluate it through a 90s test. The main indicators of concern are the amount of correctly completed conversions within 90s and the maximum continuous number of correctly completed conversions.
The Stroop color test | baseline, 1 and 2 years after follow-up
  The changes in The Stroop color test will constitute the secondary research outcome measure.The Stroop color word test was developed by Stroop in 1935 and is used to evaluate the attention function of the subject. The subject is required to correctly read the target color on the stimulus card and record the completion time. The final completion time is the score of the participant. The shorter the time used, the better the performance of the subjects
CTT (Color Trail Test) | baseline, 1 and 2 years after follow-up
  The changes in CTT will constitute the secondary research outcome. The Color Trail Test (CTT) is divided into two parts, part A and part B. Part A requires the subject to connect 25 Numbers on the paper in sequence, and part B requires the subject to connect 25 Numbers of different colors alternately in sequence. The time it takes for the subject to complete all the Numbers is the subject's final score.In this study, the investigators suspect that scores would decrease after follow-up.
ROCF (Rey-Osterrieth Complex Figure) | baseline, 1 and 2 years after follow-up
  The changes in The Rey-Osterrieth complex figure will constitute the secondary research outcome measure. The Rey-Osterrieth Complex Figure Test (ROCF), which was developed by Rey in 1941 and standardized by Osterrieth in 1944, is a widely used neuropsychological test for the evaluation of visuospatial constructional ability and visual memory. At the first step, subjects are given the ROCF stimulus card, and then asked to draw the same figure. Subsequently, they are instructed to draw what they remembered within 10 minutes. Finally, score according to the unified standard.
JoLO (Judgment of Line Orientation) | baseline, 1 and 2 years after follow-up
  The changes in Judgment of Line Orientation will constitute the secondary research outcome measure. The Judgment of Line Orientation (JLO) test is one of the most widely used measures for the assessment of visuospatial perception, and is often used for visuospatial defects after right hemisphere injury.
VFT (Verbal Fluency Test) | baseline, 1 and 2 years after follow-up
  The changes in The Verbal Fluency Test (VFT) will constitute the secondary research outcome measure. The VFT can be used to evaluate the frontal lobe fluency of patients, mainly including semantic verbal fluency and phonemic verbal fluency.
BNT (Boston Naming Test) | baseline, 1 and 2 years after follow-up
  The changes in The Verbal Fluency Test (VFT) will constitute the secondary research outcome measure. The VFT can be used to evaluate the frontal lobe fluency of patients, mainly including semantic verbal fluency and phonemic verbal fluency.
LANT (Lateralized attention network test) | baseline, 1 and 2 years after follow-up
  Attention is an important part of human cognitive function. The vigilant attention network, directed attention network and executive function network in bilateral cerebral hemispheres of asymptomatic ICAS patients can be measured by LANT.
HAMD (Hamilton Depression Scale) | baseline, 1 and 2 years after follow-up
  The changes in HAMD will constitute the secondary research outcome. Hamilton Depression Scale (HAMD) compiled by Hamilton in 1960, is the most common clinical to assess Depression Scale. In this study, 17 versions were selected, and there were 17 questions. The subjects were assessed for their depression in the past week. Each question scored between 0 and 4 points.Higher scores indicate more depressive symptoms.
HAMA (Hamilton Anxiety Scale) | baseline, 1 and 2 years after follow-up
  The changes in HAMA will constitute the secondary research outcome. Hamilton Anxiety Scale (HAMA) was compiled by Hamilton in 1959.It was one of the most commonly used scales in psychiatric clinic, including 14 items. It is often used in clinical diagnosis and degree classification of anxiety disorder. The subjects were assessed for their anxiety in the past week. Each question scored between 0 and 4 points. The higher the score, the more symptoms of anxiety.
MRI measure- resting state MRI images | baseline, 1 and 2 years after follow-up
  The resting state magnetic resonance data were collected to compare the neuroimaging differences between the patients and healthy control groups.
MRI measures-structural phase MRI images | baseline, 1 and 2 years after follow-up
  The structural phase magnetic resonance data were collected to compare the neuroimaging differences between the patients and healthy control groups.
MRI measures-3D pCASL images | baseline, 1 and 2 years after follow-up
  The three-dimensional pseudo continuous Arterial Spin Labeling (3D pCASL) data were collected to compare the differences in cerebral perfusion between the patients and healthy control groups.
Ultrasound measures-MCA-PI(middle cerebral artery-pulsatility index) | baseline, 1 and 2 years after follow-up
  Pulsatility index (PI) in the middle cerebral artery (MCA) is considered a measure of peripheral vascular resistance. The investigators want to explore the peripheral vascular resistance by MCA-PI.
Ultrasound measures-IMT( intima-media thickness) | baseline, 1 and 2 years after follow-up
  The carotid intima-media thickness (IMT) is a widely used surrogate marker for atherosclerosis worldwide. The investigators want to explore the risk of recurrence of cerebrovascular events by IMT.
Ultrasound measures-BHI(breath-holding index) | baseline, 1 and 2 years after follow-up
  The breath-holding index (BHI) is a useful method to assess cerebrovascular reactivity. The investigators want to explore the possible relationship between cognitive function and cerebrovascular reactivity by BHI.
Blood Metabolomics measures-CRP(C-reactive protiein) | baseline, 1 and 2 years after follow-up
  CRP is a plasma protein synthesized by the liver and is often used as a nonspecific biomarker of inflammation. Elevated CRP levels are associated with increased risk of cerebrovascular disease and dementia. The investigators intend to use CRP to explore the relationship between inflammatory response and cognitive impairment.
Blood Metabolomics measures-oxLDL(Oxidized low-density lipoprotein) | baseline, 1 and 2 years after follow-up
  Oxidized low-density lipoprotein (oxLDL) is a biomarker that is a key factor for the occurrence and development of atherosclerosis and the formation of unstable plaque. Atherosclerosis has been associated with the onset, severity and progression of cognitive dysfunction. The investigators intend to further explore the relationship between LDL level and cognitive impairment.
Blood Metabolomics measures-miRNA（microRNA） | baseline, 1 and 2 years after follow-up
  microRNA (miRNA) is a type of non-coding single-stranded small RNA that plays a role in biological functions by regulating post-transcriptional gene expression. miRNA is involved in the regulation of synaptic plasticity and is related to learning and memory. The investigators intend to reserve serum samples for the study of miRNA and cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China